CLINICAL TRIAL: NCT05115084
Title: The Effect of the COVID-19 Epidemic Process on the Nutritional Habits and Body Weights of Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gülin Öztürk Özkan, Associate professor, Istanbul Medeniyet University
Other Study IDs: 2021/23
Record Dates: First submitted 2021-11-06; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Pandemic; Eating Habit; Weight Gain
MeSH Terms: conditions — COVID-19; Feeding Behavior; Weight Gain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
During the COVID-19 epidemic, the time spent by adults on the stomach has increased. Therefore, the likelihood of adverse changes in lifestyles has increased. In this study, the changes in nutritional habits, physical activities and body weights of adult individuals during the epidemic will be evaluated. A questionnaire including questions about nutritional habits, physical activity status and changes in body weights will be administered to individuals. The results will be evaluated with the appropriate statistical method. The survey will be administered once. The estimated time to reach the total number is 3 months.

ELIGIBILITY:
Inclusion Criteria: Adult individuals wishing to participate in the study -

Exclusion Criteria: Individuals outside the age range of 19-70 years, all individuals who did not agree to participate in the study.

-

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals between the ages of 19 and 70 who agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-12-03 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-02 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 12 weeks
  A questionnaire containing a total of 45 questions will be applied, of which 10 are for demographic information, 31 for determining changes in body weight and eating habits, and 4 for physical activity.